CLINICAL TRIAL: NCT05807451
Title: Anatomic Relationship Of the Popliteal Vessels In Two Types Of Open Wedge High Tibial Osteotomy ( Monoplanar VS Biplanar )
Brief Title: Anatomic Relationship Of the Popliteal Vessels In Open Wedge Osteotomy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Ayman Farouk, Principal Investigator, Assiut University
Other Study IDs: Tibial Osteotomy
Record Dates: First submitted 2022-08-09; First posted 2023-04-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monoplanar Osteotomy group: High Tibial Osteotomy using single plane osteotomy
  Interventions: Procedure: High Tibial Osteotomy (Uniplanar and Biplanar )
- Biplanar Osteotomy group: High Tibial Osteotomy using two plane osteotomy
  Interventions: Procedure: High Tibial Osteotomy (Uniplanar and Biplanar )

INTERVENTIONS:
Procedure: High Tibial Osteotomy (Uniplanar and Biplanar ) — High Tibial Osteotomy using monoplanar and biplanar osteotomy techniques

SUMMARY:
The Aim Is To Study The Anatomic Relationship Of The Popliteal Vesseles In Two Types Of (OWHTO) Techniques (Monoplanar VS Biplanar) Which Provide More Safe Technique To The PV

DETAILED DESCRIPTION:
Open wedge High tibial osteotomy (OWHTO) is a common surgical Procedure that is utilized to correct knee varus deformity and prevent development or advancement of medial compatment knee osteoarthritis.

By turning the mechanical weight-bearing axis to the lateral side it correct lower limb alignment,decrease medial compartment load,pain,arthritic changes, postpone the need for arthroplasty and allow cartilage regeneration.

Like any other surgical procedure (OWHTO) has its own complications.injury to the popliteal vessels (PV) is catastrophic and limb threatening compliation that had been reported with prevalence rate ranging from 0.4% to 1.7% PV runs close to the posterior tibial cortex it might be injured while taking osteotomy cut. To avoid this problem many studies with different tools done to define PV position and its relations to provide safe technique for osteotomy.

(OWHTO) has different methods: Monoplanar and Biplanar osteotomy are most popular,both techniques differ in cut level and shape.

In this study the investigators compare between the two methods (Monoplanar VS Biplanar) concerning their proximity and safety to the PV .

Our hypothesis is that there is increase in the distance between the PV and the posterior tibial cortex the more distal the osteotomy level.

Previous studies cadaveric or preoperative studies provide useful informations with some different results , to the best of our knowledge postoperative studies rarely reported in this subject , the investigators hope this study could provide valuable informations,recommend safer technique and improve surgical outcomes from this procedure.

ELIGIBILITY:
Inclusion Criteria:

* age 30-60
* BMI less than 40
* isolated medial compartment OA
* mild to moderate degree OA Grade 2 to 3 according to kellgren&Lawrence classification
* near normal lateral and patellofemoral compartment
* intact lateral meniscus
* varus malalignment less than 15 degree
* functional range of motion

Exclusion Criteria:

* inflammatory arthritis
* post traumatic arthritis
* patients with previous peripheral arterial injury
* disease or prior insertion of metallic stent in the PV
* patient allergic to contrast agent
* patient with renal impairement
* Patients who refuse to participate in the study
* Patients who are not available for follow up

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient Of Assuit univeristy hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
comparing between (OWHTO) methods Monoplanar and Biplanar which provide more safe technique to the PV. | 3 months
  measuring distance (in mm) between Popliteal Vessels and Posterior Tibial Cortex at each osteotomy level using CT Angiography

SECONDARY OUTCOMES:
pain and function using Oxford Knee Score | 6 month
  patient reports outcome questionnaire pre and post operative,measuring patient satisfaction,the score range from 0 to 48 (the higher the better the outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Hesham El Kady, Professor, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Amendola A, Bonasia DE. Results of high tibial osteotomy: review of the literature. Int Orthop. 2010 Feb;34(2):155-60. doi: 10.1007/s00264-009-0889-8. Epub 2009 Oct 17. PMID 19838706
- [Background] Sabzevari S, Ebrahimpour A, Roudi MK, Kachooei AR. High Tibial Osteotomy: A Systematic Review and Current Concept. Arch Bone Jt Surg. 2016 Jun;4(3):204-12. PMID 27517063
- [Background] Kanamiya T, Naito M, Hara M, Yoshimura I. The influences of biomechanical factors on cartilage regeneration after high tibial osteotomy for knees with medial compartment osteoarthritis: clinical and arthroscopic observations. Arthroscopy. 2002 Sep;18(7):725-9. doi: 10.1053/jars.2002.35258. PMID 12209429
- [Background] Coventry MB. Upper tibial osteotomy. Clin Orthop Relat Res. 1984 Jan-Feb;(182):46-52. PMID 6692627
- [Background] Woodacre T, Ricketts M, Evans JT, Pavlou G, Schranz P, Hockings M, Toms A. Complications associated with opening wedge high tibial osteotomy--A review of the literature and of 15 years of experience. Knee. 2016 Mar;23(2):276-82. doi: 10.1016/j.knee.2015.09.018. Epub 2015 Nov 17. PMID 26596554
- [Background] Attinger MC, Behrend H, Jost B. Complete rupture of the popliteal artery complicating high tibial osteotomy. J Orthop. 2014 Oct 3;11(4):192-6. doi: 10.1016/j.jor.2014.08.002. eCollection 2014 Dec. PMID 25561756
- [Background] Chun KC, So BJ, Kang HT, Chun CH. Pseudoaneurysm Formation due to Popliteal Artery Injury Caused by Drilling during Medial Opening Wedge High Tibial Osteotomy. Knee Surg Relat Res. 2018 Dec 1;30(4):364-368. doi: 10.5792/ksrr.18.039. PMID 30466257
- [Background] Mori A, Matsushita T, Miyaji N, Nagai K, Araki D, Kanzaki N, Matsumoto T, Niikura T, Hoshino Y, Kuroda R. Analysis of popliteal artery location for high tibial and distal tuberosity osteotomy using contrast-enhanced computed tomography. Knee Surg Relat Res. 2022 May 8;34(1):25. doi: 10.1186/s43019-022-00154-2. PMID 35527280
- [Background] Kim J, Allaire R, Harner CD. Vascular safety during high tibial osteotomy: a cadaveric angiographic study. Am J Sports Med. 2010 Apr;38(4):810-5. doi: 10.1177/0363546510363664. Epub 2010 Mar 3. PMID 20200321
- [Background] Lee YS, Lee BK, Kim WS, Choi JS, Baek JR, Moon CW. Sagittal and coronal plane location of the popliteal artery in the open-wedge high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2014 Nov;22(11):2629-34. doi: 10.1007/s00167-013-2503-2. Epub 2013 Apr 17. PMID 23592027
- [Background] Kang T, Lee DW, Park JY, Han HS, Lee MC, Ro DH. Sawing toward the fibular head during open-wedge high tibial osteotomy carries the risk of popliteal artery injury. Knee Surg Sports Traumatol Arthrosc. 2020 May;28(5):1365-1371. doi: 10.1007/s00167-019-05439-w. Epub 2019 Feb 26. PMID 30809721
- [Background] Lobenhoffer P, Agneskirchner JD. Improvements in surgical technique of valgus high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2003 May;11(3):132-8. doi: 10.1007/s00167-002-0334-7. Epub 2003 Jan 11. PMID 12774149
- [Background] Choi CH, Lee WS, Jung M, Moon HS, Lee YH, Oh J, Kim SJ, Kim SH. Adequate protection rather than knee flexion prevents popliteal vascular injury during high tibial osteotomy: analysis of three-dimensional knee models in relation to knee flexion and osteotomy techniques. Knee Surg Sports Traumatol Arthrosc. 2020 May;28(5):1425-1435. doi: 10.1007/s00167-019-05515-1. Epub 2019 May 22. PMID 31119339